CLINICAL TRIAL: NCT06630273
Title: Canadian Initiative to Measure, Predict and Assess Cancer Treatment Outcomes in Patients Treated With Immuno-Oncotherapeutics
Acronym: (CAN-IMPACT-IO
Status: Not yet recruiting | Type: Observational
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Other Study IDs: PM2
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A fresh tumour biopsy with up to 6 cores of tumour
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrollment: Correlative Collection until time of disease progression of protocol specific IO therapy

SUMMARY:
The researchers doing this study are interested in doing the following:

* Biomarker research using fresh tumour tissue and normal blood cells, and if required, tumour tissue already collected.
* Bio-banking for use in future research using the collected tumour tissue / blood .

DETAILED DESCRIPTION:
This study is being done to enable the collection and study of these samples. The results will also look at information on how participants with this type of cancer who received immunotherapy responded to treatment.

Bio-banking is the collection, storage, and use of human body samples and related health information for future research. It provides an important resource for health research locally, across Canada, and around the world. The researchers doing the main study also are interested in storing any left-over tissue and/or blood samples that have not been used up for future research. The research that may be done on these samples in the future is unknown at this time.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to submit a blood sample for buffy-coat and at least one tumour biospecimen.
* CAN-PREDICT-IO subgroup:

Provision of pre-treatment fresh tumour biopsy/resection tumour tissue for patients who will receive IO treatment, in a specified list of IO therapeutic trials currently active in CCTG.

OR

* CAN-PIVOT subgroup:

Provision of on-treatment or at-progression fresh tumour biopsy/resection tumour tissue for patients who have received IO treatment, in a specified list of IO therapeutic trials currently active in CCTG.

There are 2 CAN-PIVOT subgroups: Primary resistance is defined as disease progression evident in initial on-treatment imaging or disease stability lasting less than six months. Acquired resistance, on the other hand, manifests as disease progression subsequent to an initial partial or complete response or after a period of disease stability lasting six months or more. Patients on adjuvant treatment, with no evidence of disease (NED) by radiological assessment who develop disease (local recurrence or metastases) after or while on immunotherapy are included.

* Archived formalin fixed paraffin embedded (FFPE) blocks or slides would only be collected from patients who met CAN-IMPACT-IO study criteria and underwent fresh tumour biopsy/resection following consent but had a tumour specimen deemed insufficient for WGTS. The FFPE sample may be used to provide an alternate source of tumour tissue for WGTS in such cases. Where local centre regulations prohibit submission of blocks of tumour tissue, a predetermined number of unstained slides of representative tumour tissue may substitute the tumour block.
* Participant consent for the CAN-IMPACT-IO study must be appropriately obtained in accordance with applicable local and regulatory requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in a specified list of immuno-oncology (IO) therapeutic trials with immune checkpoint inhibitors targeting PD1/PDL1 as single agents or in combination currently active in CCTG.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of a diverse bank of biological samples, stem cell lines, derivatives, and associated information. | 3 years
  There are no primary endpoints planned for this biobank; endpoints will be specific to research projects that utilize samples/data contained in the biobank. Projects may investigate the biology , etiology, manifestations, progression, risk factors, genetic underpinnings, and treatment of diseases, conditions, and traits.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, Study Chair — University Health Network, Princess Margaret Cancer Centre, Toronto, ON Canada; Anna Spreafico, Study Chair — University Health Network, Princess Margaret Cancer Centre, Toronto, ON Canada

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG policy
URL: https://www.ctg.queensu.ca/public/policies